CLINICAL TRIAL: NCT00447278
Title: A Randomized, Controlled, Open-Label Study of the Long-Term Impact on Functioning Using Atomoxetine Hydrochloride Compared to Other Early Standard Care in the Treatment of Attention-Deficit/Hyperactivity Disorder in Treatment-Naïve Children and Adolescents
Brief Title: A Study Comparing the Effect of Atomoxetine Versus Other Standard Care Therapy on the Long Term Functioning in Attention-Deficit/Hyperactivity Disorder (ADHD) Children and Adolescents
Acronym: ADHD LIFE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11576; B4Z-EW-LYDY (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Results first posted 2010-04-20 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

ARMS (2):
- Atomoxetine (Experimental): 0.5 mg/kg/day once a day (QD) or twice a day (BID) for 1 week then 1.2-1.8 mg/kg/day QD or BID for 6 months, up to an additional 6 months optional extension
  Interventions: Drug: Atomoxetine
- OEST (Active Comparator): Other Early Standard Treatment (OEST): any treatment for ADHD as prescribed by investigator, 6 months, up to an additional 6 months extension
  Interventions: Drug: Other standard therapy for ADHD

INTERVENTIONS:
Drug: Atomoxetine — 0.5 mg/kg/day once a day (QD) or twice a day (BID) for 1 week then 1.2-1.8 mg/kg/day QD or BID for 6 months, up to an additional 6 months optional extension
  Other Names: LY139603; Strattera
  Arms: Atomoxetine
Drug: Other standard therapy for ADHD — Any treatment for ADHD as prescribed by investigator, 6 months, up to an additional 6 months extension
  Arms: OEST

SUMMARY:
The purpose of this study is to demonstrate that atomoxetine is superior to other early standard therapy (any treatment that investigator considers is appropriate to initiate for the treatment of Attention-Deficit/Hyperactivity Disorder [ADHD]) on the long term functioning in approximately 400 children and adolescents with ADHD. Patients will be pharmacological naïve prior to entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * 6 to 16 years old
  * Diagnosis of ADHD according to Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM IV) confirmed by Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children-Present and Lifetime Version (SADS PL)
  * Pharmacological naïve
  * Normal intelligence as assessed by investigator
  * Each patient (and/or legally authorized patient representative where required by local law) must understand the nature of the study and must sign an Informed Consent Document.

Exclusion Criteria:

* Exclusion criteria

  * History of bipolar disorder, any history of psychosis or autism spectrum disorder
  * History of any seizure disorder
  * Significant prior or current medical conditions
  * History of alcohol or drug abuse within the past 3 months
  * Patients who are taking concurrently any of the excluded medications in the study.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 399 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoboken
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amiens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Ireland (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westside, Galway
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dublin
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Messina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., S.Vito Tagliamento
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Donà di Piave
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Insurgentes Cuicuilco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma Sur
- Norway (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fredrikstad
- Spain (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donostia / San Sebastian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Espluges de Llobregat
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basildon, Essex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wigan, Lancashire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield, South Yorkshire

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of a 1 week screening (Period I); 6 months open-label (Period II); Optional additional 6 month open-label extension (Period III).
Period: Period II (6 Month Open-Label)
Arm/Group | Atomoxetine | OEST
Started | 199 | 200
Received at Least One Dose of Study Drug | 199 | 199 (1 patient withdrew due to parent/guardian decision prior to receiving study drug.)
Completed | 157 | 171
Not Completed | 42 | 29
Not completed — Adverse Event | 7 | 3
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol Violation | 10 | 7
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 4 | 1
Not completed — Lack of Efficacy | 11 | 1
Not completed — Parent/Guardian Decision | 9 | 10
Period: Period III (Optional 6 Month Extension)
Arm/Group | Atomoxetine | OEST
Started | 139 (18 choose not to enter this optional period.) | 155 (16 choose not to enter this optional period.)
Completed | 109 | 140
Not Completed | 30 | 15
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 6 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Lack of Efficacy | 4 | 0
Not completed — Parent/Guardian Decision | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | OEST | Total
Number analyzed (Participants) | 199 | 199 | 398
Age Continuous [Mean (Standard Deviation); unit: years] | 9.2 (2.57) | 9.4 (2.64) | 9.3 (2.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 158 | 158 | 316
Race/Ethnicity, Customized [Number; unit: participants]
  African | 0 | 2 | 2
  Caucasian | 180 | 181 | 361
  East Asian | 2 | 1 | 3
  Hispanic | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  France | 32 | 32 | 64
  Mexico | 11 | 12 | 23
  Belgium | 23 | 23 | 46
  Spain | 61 | 58 | 119
  Ireland | 3 | 2 | 5
  Turkey | 23 | 24 | 47
  Norway | 10 | 10 | 20
  United Kingdom | 16 | 18 | 34
  Italy | 20 | 20 | 40
Kiddie Schedule for Affective Disorders - Affective Disorder [Number; unit: participants] — The Kiddie-SADS-Present and Lifetime Version is an instrument completed through a semi-structured diagnostic interview designed to assess current and lifetime history of psychopathology in children and adolescents according to Diagnostic and Statistical Manual of Mental Disorders Third Edition, Revision (DSM-III-R) and DSM Fourth Edition (DSM-IV) criteria. The 'Summary Lifetime Diagnoses Checklist' aggregates diagnoses-related data to make a final decision as to the presence or absence of the evaluated condition/disease.
  participants
    0 Affective Disorders | 189 | 189 | 378
    1 Affective Disorder | 2 | 1 | 3
    Missing Information | 8 | 9 | 17
Kiddie Schedule for Affective Disorders - Anxiety Disorder [Number; unit: participants] — The Kiddie-SADS-Present and Lifetime Version is an instrument completed through a semi-structured diagnostic interview designed to assess current and lifetime history of psychopathology in children and adolescents according to Diagnostic and Statistical Manual of Mental Disorders Third Edition, Revision (DSM-III-R) and DSM Fourth Edition (DSM-IV) criteria. The 'Summary Lifetime Diagnoses Checklist' aggregates diagnoses-related data to make a final decision as to the presence or absence of the evaluated condition/disease.
  participants
    0 Anxiety Disorders | 176 | 173 | 349
    1 Anxiety Disorder | 11 | 18 | 29
    2 Anxiety Disorders | 4 | 6 | 10
    3 Anxiety Disorders | 2 | 0 | 2
    4 Anxiety Disorders | 1 | 0 | 1
    Missing Information | 5 | 2 | 7
Kiddie Schedule for Affective Disorders - Attention-Deficit/Hyperactivity Disorder (ADHD) Subtypes [Number; unit: participants] — The Kiddie-SADS-Present and Lifetime Version is an instrument completed through a semi-structured diagnostic interview designed to assess current and lifetime history of psychopathology in children and adolescents according to Diagnostic and Statistical Manual of Mental Disorders Third Edition, Revision (DSM-III-R) and DSM Fourth Edition (DSM-IV) criteria. The 'Summary Lifetime Diagnoses Checklist' aggregates diagnoses-related data to make a final decision as to the presence or absence of the evaluated condition/disease.
  participants
    Combined ADHD Subtype | 156 | 156 | 312
    Hyperactive/Impulsive ADHD Subtype | 4 | 7 | 11
    Inattentive ADHD Subtype | 39 | 36 | 75
Kiddie Schedule for Affective Disorders - Conduct Disorder [Number; unit: participants] — The Kiddie-SADS-Present and Lifetime Version is an instrument completed through a semi-structured diagnostic interview designed to assess current and lifetime history of psychopathology in children and adolescents according to Diagnostic and Statistical Manual of Mental Disorders Third Edition, Revision (DSM-III-R) and DSM Fourth Edition (DSM-IV) criteria. The 'Summary Lifetime Diagnoses Checklist' aggregates diagnoses-related data to make a final decision as to the presence or absence of the evaluated condition/disease.
  participants
    Yes (currently have the disorder) | 13 | 10 | 23
    Yes, but not present (had disorder in the past) | 2 | 2 | 4
    No (never had the disorder) | 184 | 187 | 371
Kiddie Schedule for Affective Disorders - Oppositional Defiant Disorder [Number; unit: participants] — The Kiddie-SADS-Present and Lifetime Version is an instrument completed through a semi-structured diagnostic interview designed to assess current and lifetime history of psychopathology in children and adolescents according to Diagnostic and Statistical Manual of Mental Disorders Third Edition, Revision (DSM-III-R) and DSM Fourth Edition (DSM-IV) criteria. The 'Summary Lifetime Diagnoses Checklist' aggregates diagnoses-related data to make a final decision as to the presence or absence of the evaluated condition/disease.
  participants
    Yes (currently have the disorder) | 79 | 73 | 152
    Yes, but not present (had disorder in the past) | 2 | 4 | 6
    No (never had the disorder) | 118 | 122 | 240
Kiddie Schedule for Affective Disorders - Tic Disorder [Number; unit: participants] — The Kiddie-SADS-Present and Lifetime Version is an instrument completed through a semi-structured diagnostic interview designed to assess current and lifetime history of psychopathology in children and adolescents according to Diagnostic and Statistical Manual of Mental Disorders Third Edition, Revision (DSM-III-R) and DSM Fourth Edition (DSM-IV) criteria. The 'Summary Lifetime Diagnoses Checklist' aggregates diagnoses-related data to make a final decision as to the presence or absence of the evaluated condition/disease.
  participants
    0 Tic Disorders | 176 | 178 | 354
    1 Tic Disorder | 13 | 14 | 27
    2 Tic Disorders | 2 | 2 | 4
    3 Tic Disorders | 3 | 3 | 6
    Missing Information | 5 | 2 | 7
Age at Onset of Attention-Deficit/Hyperactivity Disorder (ADHD) [Mean (Standard Deviation); unit: years] | 4.3 (1.88) | 4.2 (1.91) | 4.2 (1.89)
Height [Mean (Standard Deviation); unit: centimeters] | 138.8 (14.59) | 140.1 (15.71) | 139.4 (15.16)
Time Since Onset of ADHD [Mean (Standard Deviation); unit: years] | 5.0 (2.65) | 5.2 (2.97) | 5.1 (2.81)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 37.5 (14.30) | 37.6 (13.35) | 37.5 (13.82)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Month Endpoint in Child Health and Illness Profile - Child Edition, Parent Report Form (CHIP-CE PRF), Achievement Domain
Description: CHIP-CE PRF: parent rated assessment of a child's health status/level of functioning. The achievement domain describes developmentally appropriate role functioning in school and with peers. The majority of items assess frequency of activities or feelings using a 5-point response format (1=never, 5=always). Standard scores (T-scores) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Normative range is 40 to 60. Higher scores indicate better health and lower scores indicate worse health.
Time Frame: Baseline, 6 months
Population: Number of participants who received at least one dose of study drug and did not have a missing value. Results for Last Observation Carried Forward (LOCF) are included.
Measure: Mean (Standard Deviation); unit: T-Scores of units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 198 | 199
T-Scores of units on a scale
  Baseline (n=198, n=199) | 28.0 (12.04) | 28.3 (12.28)
  Change from Baseline at 6 Months (n=150, n=166) | 8.4 (10.15) | 12.4 (11.37)
  Change from Baseline: 6 Month LOCF (n=192,n=195) | 7.3 (10.71) | 11.7 (11.24)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for Change from Baseline at 6 Months. P-value is not adjusted and the threshold is 0.05; Mixed model repeated measure analysis with terms for corresponding baseline T-score, treatment, country, visit, and treatment-by-visit interaction; Least Squares Mean Difference = -4.36, 95% CI 2-sided [-6.47 to -2.25] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 2: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Change from Baseline: 6 Month LOCF; Least Squares Mean Difference = -4.60, 95% CI 2-sided [-6.56 to -2.63] — Least Squares Mean Difference = Atomoxetine minus OEST

2. Secondary Outcome: Change From Baseline to 4 Month and 12 Month Endpoints in CHIP-CE PRF, Achievement Domain
Description: as for outcome 1
Time Frame: Baseline, 4 months, 12 months
Population: Number of participants who received at least one dose of study drug and did not have a missing value. Last observation carried forward (LOCF). Change at 12 months is in the participants who continue in the optional extension period (atomoxetine n= 139, OEST n=155). Their data at 6 months was taken as baseline for the 12 month change.
Measure: Mean (Standard Deviation); unit: T-Scores of units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 198 | 199
T-Scores of units on a scale
  Change from Baseline: 4 Month LOCF (n=192, n=195) | 7.8 (10.84) | 10.7 (11.32)
  Month 6 Baseline (M6B) (n=132, n=148) | 37.7 (11.75) | 41.2 (12.28)
  Change from M6B at 12 Months (n=104, n=128) | 1.2 (10.60) | -0.9 (9.51)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Change from Baseline: 4 Month LOCF; Least Squares Mean Difference = -3.10, 95% CI 2-sided [-5.08 to -1.13] — Least Squares Mean Difference = Atomoxetine minus OEST

3. Secondary Outcome: Change From Baseline to 4 Month, 6 Month, and 12 Month Endpoints in the CHIP-CE PRF Domain Scores (Satisfaction, Comfort, Resilience and Risk Avoidance)
Description: CHIP-CE PRF: parent rated assessment of a child's health status and level of functioning. Domains: Satisfaction, Comfort, Risk Avoidance, Resilience. The majority of items assess frequency of activities or feelings using a 5-point response format (1=never, 5=always). Standard scores (T-scores) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Normative range is 40 to 60. Higher scores indicate better health and lower scores indicate worse health.
Time Frame: Baseline, 4 months, 6 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Scores of units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 199 | 199
T-Scores of units on a scale
  Comfort Baseline (n=198, n=198) | 43.4 (11.58) | 43.0 (11.27)
  Comfort Change at 4 Month LOCF (n=191, n=194) | 1.9 (10.60) | 5.2 (11.22)
  Comfort Change at 6 Month LOCF (n=191, n=194) | 2.3 (11.14) | 4.7 (11.64)
  Comfort Month 6 Baseline (n=137, n=153) | 46.5 (10.98) | 47.7 (9.78)
  Comfort Change at 12 Months (n=109, n=134) | 0.2 (10.38) | -0.5 (10.28)
  Resilience Baseline (n=199, n=197) | 37.8 (14.59) | 38.9 (12.63)
  Resilience Change at 4 Month LOCF (n=193, n=193) | 4.9 (12.19) | 3.8 (13.38)
  Resilience Change at 6 Month LOCF (n=193, n=193) | 5.0 (12.86) | 5.5 (12.99)
  Resilience Month 6 Baseline (n=136, n=152) | 44.3 (14.78) | 45.3 (14.08)
  Resilience Change at 12 Months (n=109, n=133) | -1.6 (12.38) | -0.3 (11.98)
  Risk Avoidance Baseline (n=198, n=198) | 29.7 (20.18) | 31.2 (20.14)
  Risk Avoidance Change: 4 Month LOCF (n=192, n=194) | 9.0 (13.63) | 9.3 (14.20)
  Risk Avoidance Change: 6 Month LOCF (n=192, n=194) | 8.0 (12.90) | 9.6 (15.16)
  Risk Avoidance Month 6 Baseline (n=132, n=149) | 40.1 (16.45) | 41.1 (16.23)
  Risk Avoidance Change at 12 Months (n=104, n=130) | 1.0 (10.98) | 2.2 (10.25)
  Satisfaction Baseline (n=199, n=198) | 33.4 (16.16) | 32.8 (16.29)
  Satisfaction Change at 4 Month LOCF (n=193, n=194) | 3.1 (13.53) | 6.9 (16.18)
  Satisfaction Change at 6 Month LOCF (n=193, n=194) | 4.1 (13.51) | 7.2 (15.94)
  Satisfaction Month 6 Baseline (n=138, n=153) | 39.6 (15.73) | 40.7 (16.17)
  Satisfaction Change at 12 Months (n=110, n=134) | -0.9 (14.14) | 1.0 (10.96)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value for Comfort Change at 4 Month LOCF; Least Squares Mean Difference = -3.04, 95% CI 2-sided [-4.92 to -1.15] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 2: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.031, ANCOVA — P-value for Comfort Change at 6 Month LOCF; Least Squares Mean Difference = -2.10, 95% CI 2-sided [-4.01 to -0.20] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 3: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.629, ANCOVA — P-value for Resilience Change at 4 Month LOCF; Least Squares Mean Difference = 0.55, 95% CI 2-sided [-1.68 to 2.77] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 4: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.421, ANCOVA — P-value for Resilience Change at 6 Month LOCF; Least Squares Mean Difference = -0.96, 95% CI 2-sided [-3.30 to 1.38] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 5: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.388, ANCOVA — P-value for Risk Avoidance Change: 4 Month LOCF; Least Squares Mean Difference = -1.05, 95% CI 2-sided [-3.44 to 1.34] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 6: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.059, ANCOVA — P-value for Risk Avoidance Change: 6 Month LOCF; Least Squares Mean Difference = -2.29, 95% CI 2-sided [-4.66 to 0.09] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 7: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value for Satisfaction Change at 4 Month LOCF; Least Squares Mean Difference = -3.56, 95% CI 2-sided [-6.09 to -1.04] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 8: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.027, ANCOVA — P-value for Satisfaction Change at 6 Month LOCF; Least Squares Mean Difference = -2.91, 95% CI 2-sided [-5.49 to -0.33] — Least Squares Mean Difference = Atomoxetine minus OEST

4. Secondary Outcome: Change From Baseline to 4 Month, 6 Month, and 12 Month Endpoints in Weiss Functional Impairment Rating Scale-Parent Report (WFIRS-P)
Description: The 50-item WFIRS-P rates impairment in 6 domains of functioning: home, school, self-concept, social, activities of daily living, and risk taking. Each item is rated by the parent on a 4-point Likert scale from 0 to 3 (0="never or not at all", 1="sometimes or somewhat", 2="often or much", 3="very often or very much"). Average of non-missing values were calculated for each domain as well as the Total, which combined all 6 domains; therefore each scale including total has a range of 0 (best) to 3 (worst).
Time Frame: Baseline, 4 months, 6 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 199 | 199
units on a scale
  Total Baseline (n=192, n=194) | 1.02 (0.475) | 0.96 (0.453)
  Total Change at 4 Months LOCF (n=187, n=190) | -0.30 (0.328) | -0.35 (0.357)
  Total Change at 6 Month LOCF (n=187, n=190) | -0.30 (0.333) | -0.36 (0.363)
  Total 6 Month Baseline (n=134, n=150) | 0.62 (0.356) | 0.59 (0.344)
  Total Change at 12 Months (n=103, n=126) | -0.01 (0.247) | -0.02 (0.252)
  Home Baseline (n=196, n=199) | 1.28 (0.777) | 1.19 (0.728)
  Home Change at 4 Month LOCF (n=190, n=195) | -0.40 (0.608) | -0.45 (0.591)
  Home Change at 6 Month LOCF (n=190, n=195) | -0.40 (0.590) | -0.44 (0.599)
  Home 6 Month Baseline (n=139, n=152) | 0.74 (0.592) | 0.72 (0.557)
  Home Change at 12 Months (n=109, n=131) | 0.01 (0.414) | -0.04 (0.440)
  Daily Living Baseline (n=197, n=196) | 1.06 (0.559) | 1.07 (0.519)
  Daily Living Change at 4 Month LOCF (n=191, n=192) | -0.20 (0.477) | -0.25 (0.427)
  Daily Living Change at 6 Month LOCF (n=191, n=192) | -0.20 (0.467) | -0.27 (0.427)
  Daily Living 6 Month Baseline (n=139, n=152) | 0.82 (0.445) | 0.81 (0.429)
  Daily Living Change at 12 Months (n=108, n=131) | -0.04 (0.334) | -0.03 (0.365)
  Risk Taking Baseline (n=198, n=199) | 0.51 (0.424) | 0.45 (0.383)
  Risk Taking Change at 4 Month LOCF (n=192, n=195) | -0.16 (0.277) | -0.17 (0.272)
  Risk Taking Change at 6 Month LOCF (n=192, n=195) | -0.17 (0.285) | -0.18 (0.269)
  Risk Taking 6 Month Baseline (n=139, n=151) | 0.29 (0.312) | 0.25 (0.302)
  Risk Taking Change at 12 Months (n=109, n=130) | -0.01 (0.199) | -0.02 (0.207)
  School Baseline (n=198, n=199) | 1.24 (0.592) | 1.18 (0.617)
  School Change at 4 Month LOCF (n=192, n=195) | -0.49 (0.504) | -0.57 (0.563)
  School Change at 6 Month LOCF (n=192, n=195) | -0.49 (0.523) | -0.60 (0.565)
  School 6 Month Baseline (n=138, n=152) | 0.62 (0.459) | 0.53 (0.444)
  School Change at 12 Months (n=107, n=132) | -0.03 (0.455) | -0.03 (0.389)
  Self-Concept Baseline (n=198, n=198) | 0.94 (0.787) | 0.85 (0.726)
  Self-Concept Change at 4 Month LOCF (n=192, n=194) | -0.25 (0.738) | -0.31 (0.723)
  Self-Concept Change at 6 Month LOCF (n=192, n=194) | -0.27 (0.758) | -0.32 (0.728)
  Self-Concept 6 Month Baseline (n=137, n=132) | 0.55 (0.574) | 0.50 (0.538)
  Self-Concept Change at 12 Months (n=107, n=131) | 0.02 (0.615) | 0.02 (0.529)
  Social Baseline (n=198, n=198) | 1.02 (0.661) | 0.97 (0.602)
  Social Change at 4 Month LOCF (n=192, n=194) | -0.26 (0.491) | -0.32 (0.513)
  Social Change at 6 Month LOCF (n=192, n=194) | -0.28 (0.536) | -0.30 (0.521)
  Social 6 Month Baseline (n=139, n=152) | 0.64 (0.491) | 0.67 (0.499)
  Social Change at 12 Months (n=109, n=132) | -0.02 (0.405) | -0.03 (0.371)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value for Total Change at 4 Month LOCF; Least Squares Mean Difference = 0.073, 95% CI 2-sided [0.014 to 0.131] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 2: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value for Total Change at 6 Month LOCF; Least Squares Mean Difference = 0.085, 95% CI 2-sided [0.027 to 0.143] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 3: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.063, ANCOVA — P-value for Home Change at 4 Month LOCF; Least Squares Mean Difference = 0.094, 95% CI 2-sided [-0.005 to 0.192] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 4: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.131, ANCOVA — P-value for Home Change at 6 Month LOCF; Least Squares Mean Difference = 0.075, 95% CI 2-sided [-0.022 to 0.172] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 5: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.156, ANCOVA — P-value for Daily Living Change at 4 Month LOCF; Least Squares Mean Difference = 0.052, 95% CI 2-sided [-0.020 to 0.124] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 6: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.046, ANCOVA — P-value for Daily Living Change at 6 Month LOCF; Least Squares Mean Difference = 0.072, 95% CI 2-sided [0.001 to 0.143] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 7: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.068, ANCOVA — P-value for Risk Taking Change at 4 Month LOCF; Least Squares Mean Difference = 0.040, 95% CI 2-sided [-0.003 to 0.084] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 8: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.212, ANCOVA — P-value for Risk Taking Change at 6 Month LOCF; Least Squares Mean Difference = 0.028, 95% CI 2-sided [-0.016 to 0.073] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 9: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value for School Change at 4 Month LOCF; Least Squares Mean Difference = 0.121, 95% CI 2-sided [0.034 to 0.208] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 10: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for School Change at 6 Month LOCF; Least Squares Mean Difference = 0.150, 95% CI 2-sided [0.064 to 0.236] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 11: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.034, ANCOVA — P-value for Self-Concept Change at 4 Month LOCF; Least Squares Mean Difference = 0.125, 95% CI 2-sided [0.009 to 0.240] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 12: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.040, ANCOVA — P-value for Self-Concept Change at 6 Month LOCF; Least Squares Mean Difference = 0.119, 95% CI 2-sided [0.005 to 0.233] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 13: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.042, ANCOVA — p-value for Social Change at 4 Month LOCF; Least Squares Mean Difference = 0.085, 95% CI 2-sided [0.003 to 0.166] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 14: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.271, ANCOVA — P-value for Social Change at 6 Month LOCF; Least Squares Mean Difference = 0.048, 95% CI 2-sided [-0.038 to 0.134] — Least Squares Mean Difference = Atomoxetine minus OEST

5. Secondary Outcome: Change From Baseline to 4 Month, 6 Month, and 12 Month Endpoints in Attention-Deficit/Hyperactivity Disorder Rating Scale - Parent Version: Investigator Adminitered and Scored (ADHD-RS-IV Parent:Inv)
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54. Inattention and Hyperactivity-Impulsivity subscales consisted of 9 items each, for total subcale scores ranging from 0 to 27. Higher scores are indicative of more severe symptoms.
Time Frame: Baseline, 4 months, 6 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 199 | 199
units on a scale
  Total Baseline (n=199, n=198) | 40.87 (8.674) | 40.35 (8.818)
  Total Change at 4 Month LOCF (n=193, n=194) | -18.1 (11.726) | -20.1 (11.562)
  Total Change at 6 Month LOCF (n=193, n=194) | -17.6 (11.688) | -20.3 (11.397)
  Total 6 Month Baseline (n=137, n=154) | 20.84 (10.923) | 18.62 (10.255)
  Total Change at 12 Months (n=108, n=138) | -2.35 (9.393) | -2.71 (8.998)
  Inattention Baseline (n=199, n=198) | 21.91 (4.138) | 21.55 (4.373)
  Inattention Change at 4 Month LOCF (n=193, n=194) | -9.58 (6.510) | -11.1 (6.150)
  Inattention Change at 6 Month LOCF (n=193, n=194) | -9.15 (6.544) | -11.2 (6.339)
  Inattention 6 Month Baseline (n=137, n=154) | 11.52 (5.936) | 9.51 (5.510)
  Inattention Change at 12 Months (n=108, n=139) | -1.17 (5.359) | -1.13 (5.273)
  Hyperactivity Baseline (n=199, n=198) | 18.97 (6.082) | 18.80 (6.252)
  Hyperactivity Change at 4 Month LOCF (n=193,n=194) | -8.54 (6.166) | -8.97 (6.572)
  Hyperactivity Change at 6 Month LOCF (n=193,n=194) | -8.42 (6.189) | -9.13 (6.255)
  Hyperactivity 6 Month Baseline (n=138, n=154) | 9.36 (5.972) | 9.11 (5.770)
  Hyperactivity Change at 12 Months (n=109, n=138) | -1.24 (4.965) | -1.63 (4.644)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.034, ANCOVA — P-value for Total Change at 4 Month LOCF; Least Squares Mean Difference = 2.307, 95% CI 2-sided [0.173 to 4.440] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 2: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value for Total Change at 6 Month LOCF; Least Squares Mean Difference = 3.072, 95% CI 2-sided [0.942 to 5.202] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 3: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value for Inattention Change at 4 Month LOCF; Least Squares Mean Difference = 1.721, 95% CI 2-sided [0.544 to 2.899] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 4: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Inattention Change at 6 Month LOCF; Least Squares Mean Difference = 2.269, 95% CI 2-sided [1.086 to 3.453] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 5: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.298, ANCOVA — P-value for Hyperactivity Change at 4 Month LOCF; Least Squares Mean Difference = 0.580, 95% CI 2-sided [-0.515 to 1.676] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 6: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.119, ANCOVA — P-value for Hyperactivity Change at 6 Month LOCF; Least Squares Mean Difference = 0.865, 95% CI 2-sided [-0.225 to 1.956] — Least Squares Mean Difference = Atomoxetine minus OEST

6. Secondary Outcome: Change From Baseline to 4 Month, 6 Month, and 12 Month Endpoints in Clinical Global Impression Attention-Deficit/Hyperactivity Disorder - Severity (CGI-ADHD-S)
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline, 4 months, 6 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 199 | 199
units on a scale
  Baseline (n=199, n=199) | 5.54 (0.857) | 5.45 (0.903)
  Change at 4 Month LOCF (n=199, n=199) | -1.88 (1.252) | -1.94 (1.228)
  Change at 6 Month LOCF (n=199, n=199) | -1.94 (1.351) | -2.06 (1.323)
  6 Month Baseline (n=138, n=153) | 3.21 (1.104) | 3.17 (1.229)
  Change at 12 Months (n=109, n=137) | -0.28 (1.037) | -0.57 (0.953)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.366, ANCOVA — P-value for Change at 4 Month LOCF; Least Squares Mean Difference = 0.104, 95% CI 2-sided [-0.122 to 0.329] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 2: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.165, ANCOVA — P-value for Change at 6 Month LOCF; Least Squares Mean Difference = 0.169, 95% CI 2-sided [-0.070 to 0.407] — Least Squares Mean Difference = Atomoxetine minus OEST

7. Secondary Outcome: Change From Baseline to 4 Month, 6 Month, and 12 Month Endpoints in the CHIP-CE CRF for Children (6-11 Years)
Description: CHIP-CE CRF: child rated assessment of their health status and level of functioning. Domains: Achievement, Satisfaction, Comfort, Risk Avoidance, Resilience. The majority of items assess frequency of activities or feelings using a 5-point response format (1=never, 5=always). Standard scores (T-scores) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Normative range is 40 to 60. Higher scores indicate better health and lower scores indicate worse health.
Time Frame: Baseline, 4 months, 6 months, 12 months
Population: Number of "child" participants who received at least one dose of study drug and did not have a missing value. Last observation carried forward (LOCF). Change at 12 months is in the participants who continue in the optional extension period (atomoxetine n= 112, OEST n=124). Their data at 6 months was taken as baseline for the 12 month change.
Measure: Mean (Standard Deviation); unit: T-Scores of units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 160 | 156
T-Scores of units on a scale
  Achievement Baseline (n=157, n=155) | 35.8 (14.15) | 36.5 (13.03)
  Achievement Change at 4 Month LOCF (n=139, n=135) | 4.6 (12.29) | 7.0 (12.38)
  Achievement Change at 6 Month LOCF (n=145, n=142) | 5.1 (12.82) | 8.8 (12.19)
  Achievement 6 Month Baseline (n=108, n=117) | 43.8 (13.66) | 46.3 (12.50)
  Achievement Change at 12 Months (n=87, n=105) | -0.5 (9.71) | -0.1 (11.19)
  Comfort Baseline (n=159, n=155) | 49.1 (10.39) | 48.2 (9.20)
  Comfort Change at 4 Month LOCF (n=146, n=140) | 2.8 (9.25) | 5.2 (8.74)
  Comfort Change at 6 Month LOCF (n=147, n=143) | 3.1 (9.72) | 6.3 (9.14)
  Comfort 6 Month Baseline (n=108, n=122) | 52.2 (8.43) | 54.0 (8.15)
  Comfort Change at 12 Months (n=87, n=109) | -0.0 (7.14) | 1.4 (7.07)
  Resilience Baseline (n=159, n=155) | 46.1 (12.13) | 46.0 (11.12)
  Resilience Change at 4 Month LOCF (n=146, n=140) | 1.9 (10.52) | 1.3 (11.25)
  Resilience Change at 6 Month LOCF (n=147, n=143) | 2.9 (11.08) | 2.7 (12.08)
  Resilience 6 Month Baseline (n=108, n=122) | 50.0 (10.33) | 48.7 (11.35)
  Resilience Change at 12 Months (n=87, n=109) | -1.8 (8.97) | -1.0 (9.14)
  Risk Avoidance Baseline (n=158, n=155) | 44.1 (11.81) | 44.3 (11.65)
  Risk Avoidance Change: 4 Month LOCF (n=139, n=135) | 6.2 (11.17) | 7.6 (10.02)
  Risk Avoidance Change: 6 Month LOCF (n=145, n=142) | 6.0 (10.89) | 8.9 (10.48)
  Risk Avoidance 6 Month Baseline (n=108, n=118) | 51.2 (8.61) | 53.3 (9.02)
  Risk Avoidance Change at 12 Months (n=87, n=106) | -0.6 (8.10) | -0.4 (7.30)
  Satisfaction Baseline (n=159, n=155) | 47.1 (13.50) | 45.2 (12.18)
  Satisfaction Change at 4 Month LOCF (n=146, n=140) | 0.3 (10.40) | 4.1 (12.23)
  Satisfaction Change at 6 Month LOCF (n=147, n=143) | 0.7 (10.72) | 4.9 (12.17)
  Satisfaction 6 Month Baseline (n=108, n=121) | 49.4 (11.66) | 50.1 (11.07)
  Satisfaction Change at 12 Months (n=87, n=109) | 0.4 (10.61) | 0.5 (8.91)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.054, ANCOVA — P-value for Achievement Change at 4 Month LOCF; Least Squares Mean Difference = -2.35, 95% CI 2-sided [-4.74 to 0.04] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 2: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Achievement Change at 6 Month LOCF; Least Squares Mean Difference = -3.71, 95% CI 2-sided [-6.16 to -1.26] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 3: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.033, ANCOVA — P-value for Comfort Change at 4 Month LOCF; Least Squares Mean Difference = -1.74, 95% CI 2-sided [-3.33 to -0.14] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 4: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Comfort Change at 6 Month LOCF; Least Squares Mean Difference = -2.50, 95% CI 2-sided [-4.12 to -0.88] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 5: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.623, ANCOVA — P-value for Resilience Change at 4 Month LOCF; Least Squares Mean Difference = 0.50, 95% CI 2-sided [-1.50 to 2.50] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 6: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.880, ANCOVA — P-value for Resilience Change at 6 Month LOCF; Least Squares Mean Difference = 0.16, 95% CI 2-sided [-1.96 to 2.29] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 7: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.149, ANCOVA — P-value for Risk Avoidance Change: 4 Month LOCF; Least Squares Mean Difference = -1.40, 95% CI 2-sided [-3.31 to 0.50] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 8: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Risk Avoidance Change: 6 Month LOCF; Least Squares Mean Difference = -2.78, 95% CI 2-sided [-4.58 to -0.98] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 9: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value for Satisfaction Change at 4 Month LOCF; Least Squares Mean Difference = -2.62, 95% CI 2-sided [-4.71 to -0.52] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 10: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value for Satisfaction Change at 6 Month LOCF; Least Squares Mean Difference = -3.12, 95% CI 2-sided [-5.26 to -0.98] — Least Squares Mean Difference = Atomoxetine minus OEST

8. Secondary Outcome: Change From Baseline to 4 Month, 6 Month, and 12 Month Endpoints in the CHIP-Adolescent Edition (AE) for Adolescents (>11-17 Years)
Description: CHIP-AE CRF: adolescent rated assessment of their health status and level of functioning. Domains: Achievement, Satisfaction, Comfort, Risk Avoidance, Resilience. The majority of items assess frequency of activities or feelings using a 5-point response format (1=never, 5=always). Standard scores (T-scores) were established, with all domains and subdomains having a mean score of 50 and standard deviation of 10. Normative range is 40 to 60. Higher scores indicate better health and lower scores indicate worse health.
Time Frame: Baseline, 4 months, 6 months, 12 months
Population: Number of "adolescent" participants who received at least one dose of study drug and did not have a missing value. Last observation carried forward (LOCF). Change at 12 months is in the participants who continue in the optional extension period (atomoxetine n=27, OEST n=31). Their data at 6 months was taken as baseline for the 12 month change.
Measure: Mean (Standard Deviation); unit: T-Scores of units on a scale
Arm/Group | Atomoxetine | OEST
Number analyzed (Participants) | 39 | 43
T-Scores of units on a scale
  Achievement Baseline (n=37, n=37) | 49.1 (10.63) | 49.3 (9.72)
  Achievement Change at 4 Month LOCF (n=31, n=32) | 4.9 (11.62) | 1.5 (8.33)
  Achievement Change at 6 Month LOCF (n=32, n=35) | 3.1 (11.04) | 2.3 (7.96)
  Achievement 6 Month Baseline (n=26, n=30) | 53.7 (9.89) | 52.2 (10.91)
  Achievement Change at 12 Months (n=17, n=24) | -1.8 (5.46) | -0.5 (8.48)
  Satisfaction Baseline (n=37, n=38) | 49.7 (8.68) | 49.6 (11.62)
  Satisfaction Change at 4 Month LOCF (n=31, n=34) | 2.1 (7.21) | 2.4 (6.83)
  Satisfaction Change at 6 Month LOCF (n=32, n=36) | 2.8 (7.62) | 6.3 (8.51)
  Satisfaction 6 Month Baseline (n=26, n=30) | 51.2 (10.55) | 55.4 (7.56)
  Satisfaction Change at 12 Months (n=17, n=25) | -2.6 (4.79) | -1.4 (6.79)
  Comfort Baseline (n=37, n=38) | 53.0 (9.11) | 51.6 (9.00)
  Comfort Change at 4 Month LOCF (n=31, n=33) | 1.4 (11.24) | 2.6 (7.21)
  Comfort Change at 6 Month LOCF (n=32, n=35) | 1.3 (11.87) | 4.7 (7.27)
  Comfort 6 Month Baseline (n=26, n=30) | 55.1 (7.81) | 55.8 (6.36)
  Comfort Change at 12 Months (n=17, n=25) | 2.3 (7.26) | -0.2 (5.06)
  Risk Avoidance Baseline (n=37, n=37) | 55.2 (8.10) | 54.4 (7.95)
  Risk Avoidance Change: 4 Month LOCF (n=31, n=33) | 1.3 (6.35) | 2.0 (3.56)
  Risk Avoidance Change: 6 Month LOCF (n=32, n=35) | 0.6 (6.74) | 2.8 (3.89)
  Risk Avoidance 6 Month Baseline (n=26, n=30) | 57.5 (8.46) | 57.6 (7.12)
  Risk Avoidance Change at 12 Months (n=17, n=23) | -1.2 (4.51) | 0.1 (2.68)
  Resilience Baseline (n=35, n=37) | 45.0 (9.33) | 45.4 (7.33)
  Resilience Change at 4 Month LOCF (n=29, n=33) | 0.8 (6.92) | 0.3 (5.67)
  Resilience Change at 6 Month LOCF (n=30, n=35) | -0.7 (6.14) | 1.8 (7.36)
  Resilience 6 Month Baseline (n=26, n=30) | 44.1 (7.89) | 47.9 (8.25)
  Resilience Change at 12 Months (n=17, n=24) | -1.4 (6.25) | -1.7 (7.53)
Statistical Analysis 1: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.263, ANCOVA — P-value for Achievement Change at 4 Month LOCF. Achievement was derived from the academic achievement subdomain only; Least Squares Mean Difference = 2.39, 95% CI 2-sided [-1.83 to 6.60] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 2: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.848, ANCOVA — P-value for Achievement Change at 6 Month LOCF. Achievement was derived from the academic achievement subdomain only; Least Squares Mean Difference = 0.38, 95% CI 2-sided [-3.60 to 4.36] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 3: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.895, ANCOVA — P-value for Statisfaction Change at 4 Month LOCF; Least Squares Mean Difference = -0.19, 95% CI 2-sided [-3.01 to 2.64] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 4: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.038, ANCOVA — P-value for Satisfaction Change at 6 Month LOCF; Least Squares Mean Difference = -3.20, 95% CI 2-sided [-6.22 to -0.19] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 5: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.854, ANCOVA — P-value for Comfort Change at 4 Month LOCF; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-3.59 to 2.98] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 6: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.161, ANCOVA — P-value for Comfort Change at 6 Month LOCF; Least Squares Mean Difference = -2.26, 95% CI 2-sided [-5.45 to 0.92] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 7: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.540, ANCOVA — P-value for Risk Avoidance Change: 4 Month LOCF; Least Squares Mean Difference = -0.70, 95% CI 2-sided [-2.98 to 1.58] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 8: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.106, ANCOVA — P-value for Risk Avoidance Change: 6 Month LOCF; Least Squares Mean Difference = -1.98, 95% CI 2-sided [-4.40 to 0.44] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 9: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.833, ANCOVA — P-value for Resilience Change at 4 Month LOCF; Least Squares Mean Difference = 0.30, 95% CI 2-sided [-2.49 to 3.08] — Least Squares Mean Difference = Atomoxetine minus OEST
Statistical Analysis 10: Comparison: Atomoxetine vs OEST; Test type: Superiority or Other; p = 0.110, ANCOVA — P-value for Resilience Change at 6 Month LOCF; Least Squares Mean Difference = -2.34, 95% CI 2-sided [-5.21 to 0.54] — Least Squares Mean Difference = Atomoxetine minus OEST

9. Secondary Outcome: Correlation Between CHIP-CE Parent Rated and Pooled CHIP-CE Child Rated and CHIP AE Adolescent Rated T-Scores
Description: Pearson correlation coefficients were calculated on each domain at baseline, Month 6 and Change to Month 6 between parent-rated CHIP and pooled patient-rated (child and adolescent) CHIP.
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least one dose of study drug and had non-missing values.
Measure: Number; unit: correlation coefficient
Groups:
- Pearson Correlation Coefficient: Correlation Coefficient between parent-rated and patient-rated CHIP T-score domains.
Arm/Group | Pearson Correlation Coefficient
Number analyzed (Participants) | 398
correlation coefficient
  Achievement Baseline | 0.288
  Achievement Month 6 | 0.329
  Achievement Change to Month 6 | 0.167
  Comfort Baseline | 0.306
  Comfort Month 6 | 0.373
  Comfort Change to Month 6 | 0.286
  Resilience Baseline | 0.271
  Resilience Month 6 | 0.429
  Resilience Change to Month 6 | 0.113
  Risk Avoidance Baseline | 0.429
  Risk Avoidance Month 6 | 0.450
  Risk Avoidance Change to Month 6 | 0.296
  Satisfaction Baseline | 0.310
  Satisfaction Month 6 | 0.336
  Satisfaction Change to Month 6 | 0.133

ADVERSE EVENTS:
Time Frame: Baseline to 6 months (Study Period II)
Description: Includes all patients in Study Period II who received at least one dose of study drug.
Arm/Group | Atomoxetine | OEST
Serious Adverse Events (participants affected / at risk) | 2/199 | 2/199
Other Adverse Events (participants affected / at risk) | 150/199 | 146/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=199) | OEST (N=199)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=199) | OEST (N=199)
Abdominal pain (Gastrointestinal disorders) | 29 (40) | 22 (27)
Abdominal pain upper (Gastrointestinal disorders) | 18 (21) | 13 (13)
Nausea (Gastrointestinal disorders) | 25 (25) | 14 (14)
Vomiting (Gastrointestinal disorders) | 21 (25) | 11 (11)
Fatigue (General disorders) | 23 (24) | 5 (5)
Irritability (General disorders) | 3 (3) | 13 (13)
Nasopharyngitis (Infections and infestations) | 11 (13) | 12 (16)
Weight decreased (Investigations) | 17 (17) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 40 (40) | 50 (54)
Decreased appetite (Metabolism and nutrition disorders) | 25 (25) | 28 (29)
Headache (Nervous system disorders) | 48 (57) | 44 (56)
Somnolence (Nervous system disorders) | 13 (13) | 2 (2)
Initial insomnia (Psychiatric disorders) | 3 (3) | 11 (11)
Insomnia (Psychiatric disorders) | 4 (4) | 25 (25)
Tic (Psychiatric disorders) | 4 (4) | 10 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days